CLINICAL TRIAL: NCT05130411
Title: An Exploratory Investigation to Identify if Dame Product's "DLM" Works to Improve Sexual Desire and Mood in Females
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dame Products, Inc. (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20217-Dame
Record Dates: First submitted 2021-11-02; First posted 2021-11-23 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2022-01

CONDITIONS: Sexual Desire Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DLM - Test product (Experimental): The dietary supplement is designed to be taken in servings of two gummies per day.
  Interventions: Dietary Supplement: DLM - Test product

INTERVENTIONS:
Dietary Supplement: DLM - Test product — The group will receive 60 gummies each (to take two gummies per day) across a four-week period. Each participant shall take two gummies per day

SUMMARY:
This is a single-group, non-randomized, non-controlled, open-label observational trial to study and evaluate the efficacy of a commercial dietary supplement, called "DLM" ("test product"). It is hypothesized that the test product, which is designed as an edible gummy, will present a favorable result to increase sexual desire and improve mood.

ELIGIBILITY:
Inclusion Criteria:

* Females between 24-65 of age
* Must be in good health (don't report any medical conditions asked in the screening questionnaire)
* Experience sexuality-related personal distress (established in an online-screening questionnaire)
* Experience a regular menstrual cycle
* In the subject's opinion, previously experienced "normal sexual desire"
* Self-reported stress in their daily lives
* My present with self-reported anxiety
* Trouble being present in the moment
* Consider themselves as being busy all the time

Exclusion Criteria:

* Current urinary or vaginal infection
* Vaginal prolapse and any other disease that could interfere with the study conduction and participation
* Diagnosis of depression
* Diagnosis of anxiety
* Currently experiencing significant symptoms of a mental disorder that might interfere with study participation (e.g. eating disorder, obsessive-compulsive disorder, posttraumatic stress syndrome, bipolar disorder)
* Current substance abuse disorder
* Diagnosis of an autoimmune disease, such as multiples sclerosis and rheumatoid arthritis
* Self-reported or diagnosed hypotension (BP < 90 over 60)
* Is currently using, or has used any of the following types of medication within 6 months of screening:

Any for of antidepressants; Mood stabilizers Benzodiazepines ("tranquillizers") Cognitive enhancers or stimulants (e.g. Adderall) The following contraception: Hormonal combination birth control pill; hormonal progesterone-only birth control pill; birth control patch; NuvaRing; Nexplanon Taking insulin or other diabetes medication

* Currently, or in the past 6 months, undergoing hormone therapy
* Any medical condition that is unstable or uncontrolled
* A history of sexual trauma or abuse
* Females that are pregnant, want to become pregnant for the duration of the study, or who are breastfeeding

Ages: 24 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Born as female
Enrollment: 55 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Increase in sexual desire in women and associated improvements of mood and quality of life. [Time Frame: Baseline to 4 weeks) | 4 weeks
  Survey-based assessment (0-5 scale with 0 being the lowest possible score and 5 being the highest) of changes in sexual desire, mood, and quality of life between baseline and study intervention period.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
Undecided